CLINICAL TRIAL: NCT02245581
Title: Evaluations of Optimizing Perioperative Fluid Management on Postoperative Pain Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Yuan-Yi Chia, anesthesia doctor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS-102-036
Record Dates: First submitted 2014-09-10; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Patients Major Laminectomy Surgery

ARMS (2):
- SVV-guided fluid management (Active Comparator): SVV : Stoke volume variation
  Interventions: Procedure: SVV-guided fluid management
- CVP-guided fluid management (Active Comparator): CVP : Central venous pressure
  Interventions: Procedure: CVP-guided fluid management

INTERVENTIONS:
Procedure: SVV-guided fluid management
  Arms: SVV-guided fluid management
Procedure: CVP-guided fluid management
  Arms: CVP-guided fluid management

SUMMARY:
Patient characteristics, duration of surgery, and infusion volumes will be compared between the groups. Oxygen transport and organ function will be compared Length of hospital stay, morbidity, postoperative pain intensity were compared. Continuous variables will be analyzed using the student t-test and discrete variables will be analyzed using Chi-Square test. P-value <0.05 will be considered significant, where appropriate 95% confidence intervals will be calculated. Statistical analysis will be carried out using standardize statistical programs SPSS 12.0 for windows.

ELIGIBILITY:
Inclusion Criteria:

* All patients are undergoing elective spine laminectomy

Exclusion Criteria:

* age <20 yr
* emergency surgery
* coagulopathy
* renal and hepatic dysfunction
* hyperthyroidism, and cardiac rhythm other than sinus rhythm

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Pain at rest and movement | Post-operation Day1 to Day4

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan